CLINICAL TRIAL: NCT03150446
Title: The Usefulness of Flexible Cystoscopy for Preventing Double-J Stent Malposition After Laparoscopic Ureterolithotomy
Acronym: FC-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sung Gu Kang (Other)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Sponsor-Investigator, Sung Gu Kang, Associate Professor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FC-DM 1.0
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Urinary Stones; Ureteral Calculus
Keywords: laparoscopy; ureteral catheterization
MeSH Terms: conditions — Urinary Calculi; Ureteral Calculi

STUDY DESIGN:
Intervention Model Description: From April 2009 to June 2015, 97 male patients with stones >1.8 cm in the upper ureter underwent intracorporeal double-J stenting of the ureter after laparoscopic ureterolithotomy performed by four different surgeons. The 50 participants was performed with flexible cystoscopy through the urethral route to confirm the position of the double-J stent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group using flexible cystoscopy (Experimental): 50 patients with large upper ureteral stones underwent laparoscopic ureterolithotomy with flexible cystoscopy to confirm the correct positioning of the double-J stent. After intracorporeal insertion of the double-J catheter, additional endoscopic monitoring with flexible cystoscopy was performed. The surgeon manipulating the double-J catheter used monitor A, while an assistant inserted a flexible cystoscope into the bladder through the urethral route and determined whether the double-J stent was correctly placed in the bladder using monitor B before suturing the site of ureterotomy.
  Interventions: Device: flexible cystoscopy

INTERVENTIONS:
Device: flexible cystoscopy — After intracorporeal insertion of the double-J catheter, additional endoscopic monitoring with flexible cystoscopy was performed. The surgeon manipulating the double-J catheter used monitor A, while an assistant inserted a flexible cystoscope into the bladder through the urethral route and determined whether the double-J stent was correctly placed in the bladder using monitor B before suturing the site of ureterotomy. If the stent was well-placed, the flexible cystoscope was withdrawn. If the double-J stent was not visualized in the bladder, the surgeon pushed the stent inferiorly using a laparoscopic instrument and monitor A until the stent came out through the ureteral orifice on monitor B.
  Other Names: Laparoscopic adjustment of double-J stent

SUMMARY:
The aim of this study was to evaluate the role of flexible cystoscopy in preventing malpositioning of the ureteral stent after laparoscopic ureterolithotomy in male patients.

From April 2009 to June 2015, 97 male patients with stones >1.8 cm in the upper ureter underwent intracorporeal double-J stenting of the ureter after laparoscopic ureterolithotomy performed by four different surgeons. In the last 50 patients who underwent laparoscopic ureterolithotomy flexible cystoscopy was performed through the urethral route to confirm the position of the double-J stent, while in the first 47 correct positioning of the stent was confirmed through postoperative KUB.

DETAILED DESCRIPTION:
The treatment of large upper ureteral stones is still controversial. The American Urological Association (AUA) and the European Association of Urology (EAU) recommend that laparoscopic stone removal may be considered in rare cases in which shockwave lithotripsy (SWL), ureteroscopic lithotripsy (URS), and percutaneous nephrolithotomy fail or are unlikely to be successful. In a recent meta-analysis of treatment of large proximal ureteral stones, Torricelli et al. reported that the outcomes of laparoscopic ureterolithotomy (LUL) for larger upper ureteral stones are favorable compared with those of URS, and LUL should be considered as a first-line option when flexible ureteroscopy is not available. After such surgery, many surgeons prefer placing a double-J stent, a ureteral catheter that is passed through the ureter from the kidney to the bladder. Although double-J stent placement after LUL remains controversial, many urologists believe that it may help prevent postoperative urinary leakage.

Intracorporeal double-J stenting is technically difficult, and malpositioning often occurs after surgery in clinical practice. However, the actual rate of malpositioning of stents has not been reported yet. Although clinicians use different ways to place double-J stents precisely, accurate stent placement before the closure of the ureteral incision might be difficult to confirm.

Upward malpositioning of the stent after surgery may necessitate removal of the stent using a ureteroscope. It is difficult to remove stents in the outpatient setting without anesthesia to reduce pain and discomfort, especially in male patients.

In this study, The investigators used flexible cystoscopy through the urethral route before closure of the ureteral incision to confirm that the double-J stent was placed correctly in the bladder of male patients. Upon identification of upward malpositioning of the ureteral stent, position adjustments were performed by intracorporeally manipulating the ureteral stent through the incision site of the ureter. The aim of this study was to determine the malpositioning rate and predicting factors associated with upward malpositioning of intracorporeal double-J stents after LUL and to evaluate the usefulness of flexible cystoscopy in preventing such malpositioning in male patients.

ELIGIBILITY:
Inclusion Criteria:

* the patients with large stones (>1.8 cm in size) of the upper ureter
* male patients

Exclusion Criteria:

* the patients planing to be treated with other treatment except laparoscopic ureterolithotomy about the upper ureter stone
* female patients
* non operable patients

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
upward malpositioning of ureteral stents | 5 minutes
  whether the double-J stent was correctly placed in the bladder

CONTACTS AND LOCATIONS:
Overall Officials: Sung Gu Kang, Professor, Study Director — Department of Urology, Korea University College of Medicine
Locations (1):
- Department of Urology, Korea University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Kang SH, Cheon J, Lee JG, Kim JJ, Kang SG. The usefulness of flexible cystoscopy for preventing double-J stent malposition after laparoscopic ureterolithotomy. BMC Urol. 2017 Jun 15;17(1):44. doi: 10.1186/s12894-017-0232-4. PMID 28619091